CLINICAL TRIAL: NCT05269017
Title: The Potential Therapeutic Effect of Vitamin D Nasal Drops in the Treatment of Post COVID-19 Parosmia
Brief Title: Vitamin D Nasal Drops in Post COVID-19 Parosmia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menoufia University (Other)
Responsible Party: Principal Investigator, Ahmad Mahmoud Hamdan, Principle Investigator, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1/2022 PHAR2
Record Dates: First submitted 2022-03-04; First posted 2022-03-07 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Parosmia
Keywords: Vitamin D; Olfactory dysfunction; Parosmia; Post COVID-19 Parosmia
MeSH Terms: conditions — Olfaction Disorders | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The statistician will be blinded to the patient's group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): The case group patients will receive vitamin D3 nasal drops
  Interventions: Drug: Vitamin D3
- Control group (Active Comparator): The control group will remove local corticosteroid spray
  Interventions: Drug: Budesonide nasal spray

INTERVENTIONS:
Drug: Vitamin D3 — Devarol S amp containing 200,000 units per 2 ml giving a concentration of 5,000 units per drops for four weeks
  Arms: Case group
Drug: Budesonide nasal spray — 64 µg per puff in a dose of 1 puff for each nostril twice daily for four weeks
  Arms: Control group

SUMMARY:
The current study will be a pilot study for a randomized controlled trial conducted on patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine To evaluate the effect of vitamin D nasal drops in the treatment of post COVID 19 parosmia

DETAILED DESCRIPTION:
The current study will be a pilot study for a randomized controlled trial conducted on 60 patients recruited from the outpatient clinic of the Otorhinolaryngology Department, Menoufia Faculty of Medicine after approval of the institutional review board and taking informed written consent from every patient before participation in the study.

To be included in the study, patients should be more than 18 years old, have a history of COVID 19 infection more than three months ago as confirmed by PCR test, have a post COVID parosmia, and have no history of systemic steroid administration over the last one month. History of previous nasal surgery, underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases), and hypersensitivity to Ivermectin were the exclusion criteria for this study.

Patients of the study will be randomly and equally distributed between case and control groups using block randomization methods using 4 blocks each comprising 4 patients with 6 patterns for every block one of which was selected randomly using random numbers generated by Excel program. The case group will receive a 4 week course using Devarol S amp containing 200,000 units per 2 ml giving a concentration of 5,000 units per drop. The patients will receive two drops per nostril twice daily. The Control group will receive a 4 weeks course of local steroids in the form of budesonide (64 µg per puff in a dose of 1 puff for each nostril twice daily.

Assessment protocol:

Patients of the study will be assessed before and at the end of the treatment protocol with history taking to define the inclusion and exclusion criteria. Endoscopic examination of the nasal cavity will be performed to exclude any other intranasal pathology. The degree of parosmia will be assessed using a visual analog scale before and four weeks after treatment.

Outcome measures:

Primary outcome measures will include a comparison between the pre and post treatment values of visual analog scales of parosmia, and a comparison between case and control groups regarding the post treatment results whether no improvement, partial improvement, or complete improvement. Secondary outcome measures will include assessment of the side effects of Ivermectin nasal drops among the case group.

ELIGIBILITY:
nclusion Criteria:

* Patients should be more than 18 years old,
* Patients having a history of COVID 19 infection more than three months ago as confirmed by PCR test,
* Patients having a post COVID parosmia,
* Patients having no history of systemic steroid administration over the last one month.

Exclusion Criteria:

* History of previous nasal surgery,
* Underlying systemic diseases (like diabetes mellitus, hypertension, or autoimmune diseases),
* Hypersensitivity to vitamin D3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Comparison between the pre and post treatment values | After one month of treatment
  Comparison between the pre and post-treatment values of visual analog scale values for post-COVD-19 parosmia. The values range from 0 to 10 with 10 indicating severe parosmia.
Comparison between case and control groups regarding the post treatment results | After one month of treatment
  Comparison between case and control groups regarding the post treatment results whether no improvement, partial improvement, or complete improvement

SECONDARY OUTCOMES:
Assessment of the side effects of Ivermectin nasal drops | After one month of treatment
  Assessment of the side effects of Ivermectin nasal drops among the case group

CONTACTS AND LOCATIONS:
Locations (1):
- Menoufia Faculty of Medicine, Shibīn al Kawm, Menoufia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Study data will be available on request from the authors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication of the study results
Access Criteria: On approval of the authors of the study

REFERENCES:
- [Background] Vaira LA, Salzano G, Deiana G, De Riu G. Anosmia and Ageusia: Common Findings in COVID-19 Patients. Laryngoscope. 2020 Jul;130(7):1787. doi: 10.1002/lary.28692. Epub 2020 Apr 15. PMID 32237238
- [Background] Parma V, Ohla K, Veldhuizen MG, Niv MY, Kelly CE, Bakke AJ, Cooper KW, Bouysset C, Pirastu N, Dibattista M, Kaur R, Liuzza MT, Pepino MY, Schopf V, Pereda-Loth V, Olsson SB, Gerkin RC, Rohlfs Dominguez P, Albayay J, Farruggia MC, Bhutani S, Fjaeldstad AW, Kumar R, Menini A, Bensafi M, Sandell M, Konstantinidis I, Di Pizio A, Genovese F, Ozturk L, Thomas-Danguin T, Frasnelli J, Boesveldt S, Saatci O, Saraiva LR, Lin C, Golebiowski J, Hwang LD, Ozdener MH, Guardia MD, Laudamiel C, Ritchie M, Havlicek J, Pierron D, Roura E, Navarro M, Nolden AA, Lim J, Whitcroft KL, Colquitt LR, Ferdenzi C, Brindha EV, Altundag A, Macchi A, Nunez-Parra A, Patel ZM, Fiorucci S, Philpott CM, Smith BC, Lundstrom JN, Mucignat C, Parker JK, van den Brink M, Schmuker M, Fischmeister FPS, Heinbockel T, Shields VDC, Faraji F, Santamaria E, Fredborg WEA, Morini G, Olofsson JK, Jalessi M, Karni N, D'Errico A, Alizadeh R, Pellegrino R, Meyer P, Huart C, Chen B, Soler GM, Alwashahi MK, Welge-Lussen A, Freiherr J, de Groot JHB, Klein H, Okamoto M, Singh PB, Hsieh JW; GCCR Group Author; Reed DR, Hummel T, Munger SD, Hayes JE. More Than Smell-COVID-19 Is Associated With Severe Impairment of Smell, Taste, and Chemesthesis. Chem Senses. 2020 Oct 9;45(7):609-622. doi: 10.1093/chemse/bjaa041. PMID 32564071
- [Background] Lerner DK, Garvey KL, Arrighi-Allisan AE, Filimonov A, Filip P, Shah J, Tweel B, Del Signore A, Schaberg M, Colley P, Govindaraj S, Iloreta AM. Clinical Features of Parosmia Associated With COVID-19 Infection. Laryngoscope. 2022 Mar;132(3):633-639. doi: 10.1002/lary.29982. Epub 2021 Dec 13. PMID 34870334
- [Background] Bikle DD. Vitamin D metabolism, mechanism of action, and clinical applications. Chem Biol. 2014 Mar 20;21(3):319-29. doi: 10.1016/j.chembiol.2013.12.016. Epub 2014 Feb 13. PMID 24529992
- [Background] Wobke TK, Sorg BL, Steinhilber D. Vitamin D in inflammatory diseases. Front Physiol. 2014 Jul 2;5:244. doi: 10.3389/fphys.2014.00244. eCollection 2014. PMID 25071589
- [Background] Cho SW, Zhang YL, Ko YK, Shin JM, Lee JH, Rhee CS, Kim DY. Intranasal Treatment With 1, 25-Dihydroxyvitamin D3 Alleviates Allergic Rhinitis Symptoms in a Mouse Model. Allergy Asthma Immunol Res. 2019 Mar;11(2):267-279. doi: 10.4168/aair.2019.11.2.267. PMID 30661318
- [Background] Enkhjargal B, McBride DW, Manaenko A, Reis C, Sakai Y, Tang J, Zhang JH. Intranasal administration of vitamin D attenuates blood-brain barrier disruption through endogenous upregulation of osteopontin and activation of CD44/P-gp glycosylation signaling after subarachnoid hemorrhage in rats. J Cereb Blood Flow Metab. 2017 Jul;37(7):2555-2566. doi: 10.1177/0271678X16671147. Epub 2016 Jan 1. PMID 27671249
- [Background] Gong W, Feng Y, Yan P, Li S, Yu C, Zhou X, Xu F, Zhang D, Ren X, Zhou J, Jiang Y. [Effect of nasal instillation of vitamin D3 on patient with allergic rhinitis symptoms]. Lin Chuang Er Bi Yan Hou Tou Jing Wai Ke Za Zhi. 2014 Jul;28(14):1031-3. Chinese. PMID 25330636
- [Background] Shin YH, Ha EK, Kim JH, Yon DK, Lee SW, Sim HJ, Sung M, Jee HM, Han MY. Serum vitamin D level is associated with smell dysfunction independently of aeroallergen sensitization, nasal obstruction, and the presence of allergic rhinitis in children. Pediatr Allergy Immunol. 2021 Jan;32(1):116-123. doi: 10.1111/pai.13341. Epub 2020 Oct 8. PMID 32841423